CLINICAL TRIAL: NCT03982706
Title: Examination of Focal Therapies - MRI-Fusion, HIFU, NanoKnife and Cryotherapy
Brief Title: Examination of Focal Therapies- MRI-Fusion, HIFU, NanoKnife and Cryotherapy
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0316-16-RMC
Record Dates: First submitted 2018-08-15; First posted 2019-06-11 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2018-08

CONDITIONS: Prostate Cancer
Keywords: MRI-targeted prostate biopsy; focal treatment
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MRI-US Fusion: patients undergoing MRI targeted prostate biopsy
- Focal: patients undergoing focal treatment for localized prostate cancer (HIFU, NanoKnife, Cryotherapy)

SUMMARY:
The main objective of this study is to determine whether focal-driven therapies for diagnosis and treatment of prostate cancer are preferable over current clinical methods. Different focal procedures will be examined, including magnetic resonance imaging (MRI)-target biopsy, and focal treatment as High Intensity Focused Ultrasound (HIFU), cryoablation and Nano-Knife.

DETAILED DESCRIPTION:
Men who are scheduled to undergo a focal therapy will be given patient information sheet, which explains the study in lay terms. Fully informed consent, written or verbal (by phone) will be sought and documented before collecting any research data.

The following information will be collected for all patients:

* Demographic data: date of birth, age, gender, ethnicity, Height, weight.
* Medical History: number and results of previous biopsies, previous Protein Specific Antigen (PSA) tests.

For patients who have undergone or are scheduled to undergo MRI-US FUSION biopsy, the following information will be collected:

* MRI: MRI protocol, MRI results: suspected lesions, apparent diffusion coefficient (ADC) values.
* Biopsy procedure details and results: duration and success of procedure, number of cores taken, pathological results, following treatment (if applicable).

For patients who have undergone or are scheduled to undergo HIFU or Nano-Knife or Cryotherapy the following data will be collected:

* Procedure details.
* Evaluation of success: results of following PSA test, MRI and/or prostate biopsy.

Patients undergoing HIFU, Nano-Knife or Cryotherapy will also be asked to complete two questionnaires: IPSS, a validated lower urinary tract symptom questionnaire, and IIEF, a validated erectile function questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Men who have underwent, or are scheduled to undergo a focal therapy treatment at Ramat Aviv Medical Center or Rabin Medical Center
2. Age 18-90.

Exclusion Criteria:

None.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — participant eligibility is based on gender identity.
Study Population: Men, age 18-90, which have underwent, or are scheduled to undergo, MRI-US FUSION, HIFU, NanoKnife or Cryotherapy at the Ramat Aviv Medical Center or Rabin Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-10-28 (Actual); Primary Completion 2020-06-06 (Estimated); Study Completion 2020-06-06 (Estimated)

PRIMARY OUTCOMES:
PSA change after focal therapy (HIFU, Nano-Knife and Cryotherapy) | 5 years
  PSA will be taken every 3 months during the first year after procedure, and every 6 months in the next following 4 years
Prostate cancer detection rate and clinically significant prostate cancer detection rate of MRI-US FUSION biopsy. | 5 years
  clinically significant prostate cancer is defined as Gleason 7 and above

SECONDARY OUTCOMES:
Change in urinary symptoms measured by International Prostate Symptom Score (IPSS) questioner | 5 years
  IPSS questioner is a validated tool to assess urinary symptoms. Total score is ranged 0-35. Lower values represent a better outcome.
  IPSS will be filled before the procedure, every three months during the first year and every six months during the next four years following the procedure
Change in erectile function measured by International Index of Erectile Function (IIEF-5) questioner | 5 years
  IIEF-5 questioner is a validated tool to assess erectile function in men. Total score is ranged 1-25. Higher values represent a better outcome.
  IIEF-5 will be filled before the procedure, every three months during the first year and every six months during the next four years following the procedure

CONTACTS AND LOCATIONS:
Overall Officials: David Margel, MD PhD, Principal Investigator — Rabin Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel R, Ma J, Zou Z, Jemal A. Cancer statistics, 2014. CA Cancer J Clin. 2014 Jan-Feb;64(1):9-29. doi: 10.3322/caac.21208. Epub 2014 Jan 7. PMID 24399786
- [Background] Kaplan I, Oldenburg NE, Meskell P, Blake M, Church P, Holupka EJ. Real time MRI-ultrasound image guided stereotactic prostate biopsy. Magn Reson Imaging. 2002 Apr;20(3):295-9. doi: 10.1016/s0730-725x(02)00490-3. PMID 12117612
- [Background] Brown SB, Brown EA, Walker I. The present and future role of photodynamic therapy in cancer treatment. Lancet Oncol. 2004 Aug;5(8):497-508. doi: 10.1016/S1470-2045(04)01529-3. PMID 15288239
- [Result] Klotz L, Zhang L, Lam A, Nam R, Mamedov A, Loblaw A. Clinical results of long-term follow-up of a large, active surveillance cohort with localized prostate cancer. J Clin Oncol. 2010 Jan 1;28(1):126-31. doi: 10.1200/JCO.2009.24.2180. Epub 2009 Nov 16. PMID 19917860
- [Result] Wise AM, Stamey TA, McNeal JE, Clayton JL. Morphologic and clinical significance of multifocal prostate cancers in radical prostatectomy specimens. Urology. 2002 Aug;60(2):264-9. doi: 10.1016/s0090-4295(02)01728-4. PMID 12137824
- [Result] Pinto PA, Chung PH, Rastinehad AR, Baccala AA Jr, Kruecker J, Benjamin CJ, Xu S, Yan P, Kadoury S, Chua C, Locklin JK, Turkbey B, Shih JH, Gates SP, Buckner C, Bratslavsky G, Linehan WM, Glossop ND, Choyke PL, Wood BJ. Magnetic resonance imaging/ultrasound fusion guided prostate biopsy improves cancer detection following transrectal ultrasound biopsy and correlates with multiparametric magnetic resonance imaging. J Urol. 2011 Oct;186(4):1281-5. doi: 10.1016/j.juro.2011.05.078. Epub 2011 Aug 17. PMID 21849184
- [Result] Sonn GA, Natarajan S, Margolis DJ, MacAiran M, Lieu P, Huang J, Dorey FJ, Marks LS. Targeted biopsy in the detection of prostate cancer using an office based magnetic resonance ultrasound fusion device. J Urol. 2013 Jan;189(1):86-91. doi: 10.1016/j.juro.2012.08.095. Epub 2012 Nov 14. PMID 23158413
- [Result] Shaw GL, Thomas BC, Dawson SN, Srivastava G, Vowler SL, Gnanapragasam VJ, Shah NC, Warren AY, Neal DE. Identification of pathologically insignificant prostate cancer is not accurate in unscreened men. Br J Cancer. 2014 May 13;110(10):2405-11. doi: 10.1038/bjc.2014.192. Epub 2014 Apr 10. PMID 24722183
- [Result] Barzell WE, Melamed MR, Cathcart P, Moore CM, Ahmed HU, Emberton M. Identifying candidates for active surveillance: an evaluation of the repeat biopsy strategy for men with favorable risk prostate cancer. J Urol. 2012 Sep;188(3):762-7. doi: 10.1016/j.juro.2012.04.107. Epub 2012 Jul 19. PMID 22818143
- [Result] Wysock JS, Rosenkrantz AB, Huang WC, Stifelman MD, Lepor H, Deng FM, Melamed J, Taneja SS. A prospective, blinded comparison of magnetic resonance (MR) imaging-ultrasound fusion and visual estimation in the performance of MR-targeted prostate biopsy: the PROFUS trial. Eur Urol. 2014 Aug;66(2):343-51. doi: 10.1016/j.eururo.2013.10.048. Epub 2013 Nov 8. PMID 24262102
- [Result] Kasivisvanathan V, Dufour R, Moore CM, Ahmed HU, Abd-Alazeez M, Charman SC, Freeman A, Allen C, Kirkham A, van der Meulen J, Emberton M. Transperineal magnetic resonance image targeted prostate biopsy versus transperineal template prostate biopsy in the detection of clinically significant prostate cancer. J Urol. 2013 Mar;189(3):860-6. doi: 10.1016/j.juro.2012.10.009. Epub 2012 Oct 11. PMID 23063807
- [Result] Blana A, Murat FJ, Walter B, Thuroff S, Wieland WF, Chaussy C, Gelet A. First analysis of the long-term results with transrectal HIFU in patients with localised prostate cancer. Eur Urol. 2008 Jun;53(6):1194-201. doi: 10.1016/j.eururo.2007.10.062. Epub 2007 Nov 5. PMID 17997026
- [Result] Mearini L, D'Urso L, Collura D, Nunzi E, Muto G, Porena M. High-intensity focused ultrasound for the treatment of prostate cancer: A prospective trial with long-term follow-up. Scand J Urol. 2015;49(4):267-74. doi: 10.3109/21681805.2014.988174. Epub 2014 Dec 8. PMID 25485722
- [Result] Valerio M, Dickinson L, Ali A, Ramachadran N, Donaldson I, Mccartan N, Freeman A, Ahmed HU, Emberton M. Nanoknife Electroporation Ablation Trial: A Prospective Development Study Investigating Focal Irreversible Electroporation for Localized Prostate Cancer. J Urol. 2017 Mar;197(3 Pt 1):647-654. doi: 10.1016/j.juro.2016.09.091. Epub 2016 Sep 30. PMID 27697580
- [Result] Valerio M, Dickinson L, Ali A, Ramachandran N, Donaldson I, Freeman A, Ahmed HU, Emberton M. A prospective development study investigating focal irreversible electroporation in men with localised prostate cancer: Nanoknife Electroporation Ablation Trial (NEAT). Contemp Clin Trials. 2014 Sep;39(1):57-65. doi: 10.1016/j.cct.2014.07.006. Epub 2014 Jul 26. PMID 25072507